CLINICAL TRIAL: NCT04986033
Title: Association Between Vitamin D and Perioperative Hemoglobin Levels in Patients Undergoing Off-pump Coronary Artery Bypass Graft Surgery: Role of Hepcidin
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-0707
Record Dates: First submitted 2021-07-21; First posted 2021-08-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Preoperative anemia is present in more than 50% of patients undergoing cardiac surgery, which is associated with increased risk of transfusion, increased length of stay in the intensive care unit, and increased incidence of renal failure and mortality.

To date, clinical research on perioperative anemia has been focused on finding and treating other underlying causes of anemia, lowering the threshold for transfusion, and performing careful transfusion.

However, recently, it was known that hepcidin and erythroferrone are related to iron metabolism and absorption, vitamin D has an inverse correlation with the development of anemia, and is related to hepcidin concentration control.

Therefore, in this study, the relationship between vitamin D, hepcidin concentration and perioperative hemoglobin level in patients with off-pump coronary artery bypass graft surgery was investigated together.

ELIGIBILITY:
Inclusion Criteria:

1. Patients over 20 years of age undergoing off-pump coronary artery bypass graft

Exclusion Criteria:

1. Emergency operation
2. Minimal invasive coronary artery bypass graft
3. Cooperative operation with other surgery
4. Patients who need a mechanical ventricular assist device
5. Patients with chronic kidney disease (eGFR < 30)
6. Patients who have a end stage renal disease and need a hemodialysis
7. Patients with a low hemoglobin (Hb < 10) before surgery
8. Patients who have a some disease(leukemia, myeloma, aplastic anemia, sickle cell anemia, etc) affecting hematopoiesis
9. Patients with a liver cirrhosis
10. Patients who receive vit. D, iron supplements, erythropoietin within 6 months
11. Patients who cannot understand the informed consent (eg. Foreigner, patients with cognitive dysfunction, etc)
12. Patients who disagree this study

Min Age: 20 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who consented to study enrollment among patients scheduled for off-pump coronary artery bypass graft
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Relationship about pre-operative vitamin D level and recovery of hemoglobin | Up to 1month
  Vitamin D is a fat-soluble vitamin, a regulator acting on bone and calcium metabolism, and is known to affect the pathophysiology of several chronic diseases, and is particularly closely related to heart disease.
  Vitamin D deficiency was observed in 56% of patients undergoing cardiac surgery, and low vitamin D concentrations increased the risk of postoperative infection and organ failure, atrial fibrillation, and delirium.
  It is also known that vitamin D is closely related to anemia by regulating the secretion of erythroferrone and changing the concentration of hepcidin.

CONTACTS AND LOCATIONS:
Overall Officials: Seo Hee Ko, Principal Investigator — Division of Cardiac Anesthesiology, Department of Anesthesiology and Pain Medicine, Cardiovascular Hospital, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea
Locations (1):
- Division of Cardiac Anesthesiology, Department of Anesthesiology and Pain Medicine, Cardiovascular Hospital, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No